CLINICAL TRIAL: NCT03767647
Title: Effects of an Educational Intervention on Emotional Intelligence in School Students: Randomized Clinical Trial
Brief Title: Effects of an Educational Intervention on Emotional Intelligence in School Students
Acronym: EMCONMIGO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Severo Ochoa (Other)
Responsible Party: Principal Investigator, Blanca Navarro Peral, Nurse Resident in Mental Health, Hospital Severo Ochoa
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: pos05/18
Record Dates: First submitted 2018-12-05; First posted 2018-12-06 (Actual); Last update posted 2018-12-13 (Actual); Status verified 2018-12

CONDITIONS: Emotional Intelligence
Keywords: emotional intelligence; students; randomized clinical trial; schools

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Receives 6 lessons in 6 different weeks on Emotional Intelligence
  Interventions: Behavioral: Emotional Intelligence lessons
- Control group (No Intervention): Receives no intervention.

INTERVENTIONS:
Behavioral: Emotional Intelligence lessons — 6 lessons were given to the students in separated weeks by the same investigator. Lessons were 45-60 minutes long and each one was dedicated to one of the main aspects of emotional intelligence.
  Arms: Intervention group

SUMMARY:
Objectives: Evaluate the effect on emotional intelligence levels of an educational intervention.

Design: Randomized Clinical Trial

Methods: An intervention on emotional intelligence was conducted in a Primary School. Students were recruited and randomized into intervention or control group (no intervention) by class (cluster). Total sample was 179. Results were measured with EQi-YV and ERQ-CA questionnaires. Statistical analysis was made with Student's t and Mann-Whitney's U tests.

ELIGIBILITY:
Inclusion Criteria:

* Be on 5th or 6th year of Spanish Primary Education.
* Accept informed consent of the study.
* Be able to read, understand and answer both questionnaires

Exclusion Criteria:

* Revoque informed consent.
* Be in two different classes from the school.
* Absence to 25% or more of the lessons.
* Answer less than 80% of any questionnaire.
* Not completing both questionnaires.

Ages: 10 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 179 (Actual)
Dates: Start 2018-09-07 (Actual); Primary Completion 2018-10-22 (Actual); Study Completion 2018-10-30 (Actual)

PRIMARY OUTCOMES:
Elevation of levels of Emotional Intelligence with EQi-YV ("Emotional Quotient Inventory: youth version") questionnaire | 6 weeks
  Increment of at least 3 points of median puntuation of emotional intelligence using EQi-YV questionnaire. Range of puntuations: 60-240 points. EQi-YV is the method in Spanish with higher internal and external validity to measure emotional intelligence in children and teenager population. The participants must show their degree of agreement with 60 items on a Likert scale of 4 points (1: never happens to me, 4: it always happens to me). It consists of 5 subscales: general mood, adaptability, stress management, interpersonal skills and intrapersonal skills. All negative punctuations were positivized for analisis (5-n). Total value is obtained by the sum of the items and reflects the level of emotional intelligence. A higher value means a better condition for the patient.
Elevation of levels of Emotional Intelligence with ERQ-CA ("Emotional Regulation Questionary") questionnaire | 6 weeks
  Increment of at least 2 points of median emotional intelligence using ERQ-CA questionnaire. The ERQ-CA measures emotional regulation capacity, it has been validated in Spanish. ERQ-CA consists on 10 Likert items on a scale of 5 points (1: never happens to me; 5: it always happens to me). It is formed of two subscales: cognitive re-evaluation and emotional suppression. Total puntuation is obtained by the sum of the items and varies from 10 to 50. All negative puntuations were positivized for analisis (6-n). A higher value means a better condition for the patient.

SECONDARY OUTCOMES:
Elevation of levels of general mood subscale with EQi-YV ("Emotional Quotient Inventory: youth version") questionnaire | 6 weeks
  Increment of at least 1.5 points of median puntuation of general mood subscale using EQi-YV questionnaire. Range of puntuations 14-56. The participants must show their degree of agreement with items on a Likert scale of 4 points (1: never happens to me, 4: it always happens to me). It consists on 14 items of general mood (items 1, 4, 9, 13,19, 23, 29, 32, 37, 40, 47, 50, 56, 60). All negative punctuations were positivized for analisis (5-n). Total value represents the level of general mood. A higher value means a better condition for the patient.
Elevation of levels of adaptability subscale with EQi-YV ("Emotional Quotient Inventory: youth version") questionnaire | 6 weeks
  Increment of at least 1.5 points of median puntuation of adaptability subscale using EQi-YV questionnaire. Range of puntuations 10-40. The participants must show their degree of agreement with items on a Likert scale of 4 points (1: never happens to me, 4: it always happens to me). It consists on 10 items of adaptability (items 12, 16, 22, 25, 30, 34, 38, 44, 48, 57). All negative punctuations were positivized for analisis (5-n). Total value represents the level of adaptability. A higher value means a better condition for the patient.
Elevation of levels of stress management subscale with EQi-YV ("Emotional Quotient Inventory: youth version") questionnaire | 6 weeks
  Increment of at least 1.5 points of median puntuation of stress management subscale using EQi-YV questionnaire. Range of puntuations 12-48. The participants must show their degree of agreement with items on a Likert scale of 4 points (1: never happens to me, 4: it always happens to me). It consists on 12 items of stress management (items 3, 6, 11, 15, 21, 26, 35, 39, 46, 49, 54, 58). All negative punctuations were positivized for analisis (5-n). Total value represents the level of stress management. A higher value means a better condition for the patient.
Elevation of levels of interpersonal skills subscale with EQi-YV ("Emotional Quotient Inventory: youth version") questionnaire | 6 weeks
  Increment of at least 1.5 points of median puntuation of interpersonal skills subscale using EQi-YV questionnaire. Range of puntuations 11-44. The participants must show their degree of agreement with items on a Likert scale of 4 points (1: never happens to me, 4: it always happens to me). It consists on 11 items of interpersonal skills (items 2, 5, 10, 14, 20, 24, 36, 41, 45, 55, 59). All negative punctuations were positivized for analisis (5-n). Total value represents the level of interpersonal skills. A higher value means a better condition for the patient.
Elevation of levels of intrapersonal skills subscale with EQi-YV ("Emotional Quotient Inventory: youth version") questionnaire | 6 weeks
  Increment of at least 1.5 points of median puntuation of intrapersonal skills subscale using EQi-YV questionnaire. Range of puntuations 6-24. The participants must show their degree of agreement with items on a Likert scale of 4 points (1: never happens to me, 4: it always happens to me). It consists on 6 items of intrapersonal skills (items 7, 17, 28, 31, 43, 53). All negative punctuations were positivized for analisis (5-n). Total value represents the level of intrapersonal skills. A higher value means a better condition for the patient.
Elevation of levels of cognitive re-evaluation subscale with ERQ-CA ("Emotional Regulation Questionary") questionnaire | 6 weeks
  Increment of at least 1 point of median cognitive re-evaluation subscale using ERQ-CA questionnaire. Range of puntuations 6-30. The participants must show their degree of agreement with items on a Likert scale of 5 points (1: never happens to me; 5: it always happens to me). It consists on 6 items of cognitive re-evaluation (items 1, 3, 5, 7, 8, 10). All negative puntuations were positivized for analisis (6-n). Total value represents the level of cognitive re-evaluation. A higher value means a better condition for the patient.
Elevation of levels of emotional suppression subscale with ERQ-CA ("Emotional Regulation Questionary") questionnaire | 6 weeks
  Increment of at least 1 point of median emotional suppression subscale using ERQ-CA questionnaire. Range of puntuations 4-20. The participants must show their degree of agreement with items on a Likert scale of 5 points (1: never happens to me; 5: it always happens to me). It consists on 4 items of emotional suppression (items 2, 4, 6, 9). All negative puntuations were positivized for analisis (6-n). Total value represents the level of emotional suppression. A higher value means a better condition for the patient.

CONTACTS AND LOCATIONS:
Overall Officials: Blanca Navarro Peral, Principal Investigator — Nurse resident in Mental Health
Locations (1):
- Hospital Universitario José Germain, Leganés, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No